CLINICAL TRIAL: NCT03562273
Title: Tumor Bed Boost Using a Breast Specific Radiosurgery Device, The GammaPodTM: Registry Study and Evaluation of Quality of Life With Development of Sizing Nomogram
Brief Title: GammaPod Registry and Quality of Life Nomogram
Acronym: GCC 1876
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00080885
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female
Keywords: Breast Nomogram; Breast Cancer Quality of Life; GammaPod Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- GammaPod Quality of Life Evaluations: This study is a prospective, single arm study (registry) summarizing patient-level adverse-event and tumor outcomes as well as a number of feasibility and dosimetric characteristics of delivering a single-fraction boost with the GammaPod.
  Interventions: Radiation: Quality Of Life Sizing Nomogram

INTERVENTIONS:
Radiation: Quality Of Life Sizing Nomogram — If the participant meets the eligibility criteria of the study, and participant chooses to take part, they will receive the tumor bed boost in 8 Gy in 1 fraction just prior to starting whole breast radiation after joining the study. Treatment to the whole breast will begin within 7-8 days from the TB boost (GammaPodTM) treatment.
  The radiation therapy will take approximately 6 weeks to complete. Follow-up visits specifically for this study will continue for one year, although the physician will continue to follow as part of routine care.
  Other Names: GammaPod Quality Of Life Sizing Nomogram

SUMMARY:
This study is a prospective, single arm study (registry) summarizing patient-level adverse-event and tumor outcomes as well as a number of feasibility and dosimetric characteristics of delivering a single-fraction boost with the GammaPod.

DETAILED DESCRIPTION:
Breast conserving therapy (BCT), consisting of surgical lumpectomy followed by whole breast radiation therapy has become the standard of care for treating early-stage breast cancers. In comparison with mastectomy, BCT demonstrated similar outcomes with superior cosmesis and reduced psychological and emotional trauma based on multiple randomized trials. At the time of the lumpectomy, the surgeon removes the tumor and a surrounding rim of normal tissue (margin), typically leaving surgical clips to help designate the resection cavity or tumor bed (TB) for the radiation oncologist. The current standard of radiation therapy for breast cancer is to deliver treatment to the whole breast to 45-50.4Gy in 25 to 28 treatments Monday through Friday. Following whole breast radiation, a 'boost' is delivered to the TB in order to deliver 60 - 66Gy to the tumor bed. Two prospective trials have demonstrated a statistically significant reduction in local failures with the addition of a boost of 10Gy(in 4 fractions @ 2.5 Gy per fraction) or 16 Gy in 8 fractions @ 2 Gy per fraction), respectively.

Boost treatments can be delivered through a variety of techniques including a single electron field (used for superficial tumor beds) or multiple photon fields (2 or 3 fields typically) for tumors that are deep to the skin (usually > 3 cm). With the use of CT simulation to guide the delivery of the boost, the need for deep TB coverage has become more apparent and now most patients receive photons for the boost portion of their therapy because the use of electrons often misses part of the tumor bed. However, when photon beams are used, in comparison to electrons, more generous margins posterior to the surgical cavity are required to account for daily set up error and respiratory motion which is not necessary for a single en face electron field. Furthermore, there are only limited directions along which the radiation can be directed to the TB, and as a result, large volumes of normal breast tissue receive a substantial fraction of the prescription dose which can lead to internal scarring (fibrosis) and poor cosmesis. The largest clinical series evaluating this issue demonstrated increased fibrosis and worse cosmetic outcome using photons. The clinical target volume for the boost is the TB, while an additional 1-1.5 cm margin of normal breast tissue is added isocentrically to account for daily set-up error and respiratory motion to define a planning target volume. Typically the boost is delivered after the whole breast portion of treatment, however, in various cases this sequence can be changed. For example, if significant skin breakdown occurs during the whole breast radiation phase, investigators can stop the whole breast radiation therapy and change to deliver dose only to the TB while allowing time for the rest of the breast to heal. This allows a continuous course of therapy to the highest risk of subclinical disease (i.e. the tumor bed).

Hypofractionation, or delivery of greater than standard 1.8 - 2 Gy fraction sizes per day, is a method of shortening overall treatment time in early stage breast cancer. Historically, standard fraction sizes of 1.8-2.0 Gy for whole breast irradiation (WBI) were based primarily on studies examining squamous cell cancers from cervix and head and neck regions. The smaller fraction sizes exploited a biological differential in squamous cell cancer fractionation sensitivity versus normal tissue fractionation sensitivity. This allowed relative sparing of surrounding normal tissue from low dose per fraction. However, investigators from the United Kingdom hypothesized that the fractionation sensitivity for adenocarcinoma of the breast is close to that of the normal breast tissue. Therefore, with increasing fraction size a sufficiently large reduction of total dose could be implemented to keep late toxicity constant without reducing the probability of tumor control.

ELIGIBILITY:
Inclusion Criteria:

* The patient must sign consent for study participation.
* The patient must be female and have a diagnosis of an invasive or non-invasive breast cancer that was treated surgically by a partial mastectomy.
* The patient must be deemed an appropriate candidate for breast conserving therapy (i.e. not pregnant, never had radiation to the treated breast, breast size would allow adequate cosmesis after volume loss from partial mastectomy).
* Patients with involved lymph nodes are candidates for the study.
* Surgical margins are negative for invasive (no tumor on ink) or non-invasive breast cancer (2 mm negative margin).
* The greatest dimension of the tumor is less than 4cm before surgery.
* Multifocal disease is allowed if it was removed by a single lumpectomy resection and the patient remained a candidate for breast conservation.
* Age 18 years and older.
* Women of childbearing potential (pre-menopausal defined as having a menstrual period within the past 1 year) must have a negative serum pregnancy test or complete a pregnancy waiver form per institutional policy.
* The surgical cavity is clearly visible on CT images. Of note, clips are not required but recommended.
* The patient must weigh less than 150Kg (330lb), which is the limit of the imaging couch.
* The patient must be less than 6'6" in height.
* The patient must feel comfortable in the prone position.
* Diagnosis of prior contralateral breast cancer is allowed.
* Diagnosis of synchronous bilateral cancers is allowed. In this case if bilateral boosts are required, a patient would not have both treatments on the same day.
* Oncoplastic reduction surgery is allowed if the lumpectomy cavity can be clearly visualized.

Exclusion Criteria:

* Patients with proven multi-centric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm).
* Prior radiation therapy to that breast or that hemi thorax.
* Unable to fit into the immobilization breast cup with an adequate seal.
* Male gender.
* Patient cannot comfortably be set up in the prone position (i.e. physical disability)
* Unable to fit into the breast immobilization device due to breast size or other anatomical reason.
* Mastectomy is the surgery performed.
* Patient has received prior radiotherapy to the involved breast.
* Tumor bed is less than 3 mm from the skin surface.
* Greater than 50% of the target volume is above the upper border of the table.
* Patients with skin involvement, regardless of tumor size.
* Patients with connective tissue disorders specifically systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Patients with psychiatric or addictive disorders that would preclude obtaining informed consent.
* Patients who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females.
* Patients with breast implants/tissue expanders or flap reconstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality Of Life Evaluations | 1 year
  Evaluate the quality of life impact shortening treatment by 3-4 fractions may have on a patient via questionnaire(s).

SECONDARY OUTCOMES:
GammaPod Nomogram construction | 1 year
  Development of a sizing nomogram for the breast immobilization device using a diagram representing the relations between three or more variable quantities by means of a number of scales, so arranged that the value of one variable can be found by a simple geometric construction, for example, by drawing a straight line intersecting the other scales at the appropriate values.
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 | ~10 weeks
  Evaluate acute toxicity of the GammaPod treatment during and up to 1 month following completion of the whole breast +/- LN portion of treatment using a questionnaire.
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 post one year from treatment | ~1.5 years
  The evaluation of long-term toxicity at one year to assess the presence of subcutaneous fibrosis, and fat necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Nichols, M.D., Principal Investigator — University of Maryland
Locations (4):
- United States (4):
  - Upper Chesapeake Health, Bel Air, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland
  - UTSouthwestern, Dallas, Texas